CLINICAL TRIAL: NCT05925582
Title: Comparison of the Effects of Vestibular-based and Callisthenic-based Exercises on Cognitive Function and Dual Task in Ambulatory Older Adults Living in Nursing Homes: A Randomized Controlled Trial.
Brief Title: Vestibular-Based Exercises vs. Calisthenic Exercises for Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ugur Cavlak, Clinical Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/7614
Record Dates: First submitted 2023-06-22; First posted 2023-06-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: Two groups: Interventional (study) group and Control group
Who Masked: Participant
Masking Description: None of the participants knows the group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): All the participants in Group 1 will receive a 8-week vestibular based exercises program 3 times in a week.
  Interventions: Other: vestibular based exercise program
- Group 2 (Active Comparator): All the participants in Group 1 will receive a 8-week calistenic based exercises program 3 times in a week.
  Interventions: Other: calisthenic based exercise program

INTERVENTIONS:
Other: vestibular based exercise program — this group's participants will involve in vestibular based exercise program
  Arms: Group 1
Other: calisthenic based exercise program — this group's participants will involve in calisthenic based exercise program
  Arms: Group 2

SUMMARY:
This study was planned to determine the effects of vestibular-based exercises (VBE) and calisthenic-based exercises (CBE) on the cognitive functions of the older individuals. A total of 30 people (21 male, 9 female; range: 65 - 85) will participate in the study. In this randomized controlled study, 30 participants will be divided into two groups: VBE Group (n: 15) and CBE Group (n: 15). Standardized Mini Mental State Test (SMMT) and 3 dual task (motor + cognitive: Dual Task 1, 2, 3) tests will be used to evaluate the cognitive functions of the participants.

DETAILED DESCRIPTION:
All the evaluations will be done before and after the 8-week exercise program (three times a week). Each group participants will be divided into 3 groups (each group consists of 5 persons) and involved in an 8-week (3 days a week) exercise program (warm-up, VBE or CBE, cool-down).

ELIGIBILITY:
Inclusion Criteria:

Male and female individuals aged 65-85 years living in a nursing home.

* Individuals who are self-sufficient (independent) in daily life (including those who use a cane or canadian).
* Volunteer to participate in the study.

Exclusion Criteria:

* Having an orthopedic, neurological or psychiatric disorder that would prevent the evaluation and exercise program in the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Standardized Mini Mental State Test (SMMT) | 15 min.
  It was first developed by Folstein et al. (1975) to assess mental status. Then a standardized version was produced by Molloy and Standish (1997). The Turkish version was prepared by 3 psychiatrists (CG, TE, EE). This test, which is applied to evaluate the mental state, examines cognitive functions in five parts. These sections are; orientation, recording, attention and calculation, recall and language. The highest score is 30. Those who score 24 and below are evaluated within the framework of dementia.
Dual task 1 (Motor + Cognitive) Test | 10 min.
  Dual task 1 (Motor + Cognitive) Test This test will be used to perform a cognitive task while walking a distance of 10 meters in the person. In an area of 10 meters, the walking speed of the person is examined with the help of a stopwatch. The participant is asked to walk within a 10 meter area. Time starts when the person's foot is on the starting line and ends when he crosses the finish line. The measurement is made and the result is recorded in meters/second (m/s). In order to evaluate their cognitive functions, the participant is asked to count from 1 to 20 during walking.
Dual task 2 (Motor + Cognitive) Test | 5 min.
  The person sits down and numbers from 1 to 10 of different colors are placed on the floor. Before the test starts, 10 different commands are determined for the participant and when the test starts, these commands are said in order. The test score is determined according to the ability to execute the given commands.
Dual task 3 (Motor + Cognitive) Test | 10 min.
  Part B of the Trail Making Test will be used. The Tracking Test was first created by psychologists working in the United States Army (Reitan 1955) and is a widely used neuropsychological test. This test requires visuospatial processing and motor skills. It consists of two parts, A and B. Part A evaluates the rate of activation based on visual scanning ability, and part B evaluates the ability to change setup and follow sequencing between sets of stimuli. Part B is more complex and takes longer to complete because it requires more visual-spatial processing than part A. Also, the difficulty level of Part B is higher than Part A because it requires more motor speed, agility and attention. That's why we chose part B of the test for this research. Participants first make a short sample of the test. Then comes the actual test.

CONTACTS AND LOCATIONS:
Overall Officials: UGUR CAVLAK, Prof., Study Director — Biruni University
Locations (1):
- Faculty of Health Sciences in Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
AFTER COMPLETED THE STUDY.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2023
Access Criteria: free

REFERENCES:
- [Background] Li L, Liu M, Zeng H, Pan L. Multi-component exercise training improves the physical and cognitive function of the elderly with mild cognitive impairment: a six-month randomized controlled trial. Ann Palliat Med. 2021 Aug;10(8):8919-8929. doi: 10.21037/apm-21-1809. PMID 34488379
- [Background] Langlois F, Vu TT, Chasse K, Dupuis G, Kergoat MJ, Bherer L. Benefits of physical exercise training on cognition and quality of life in frail older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):400-4. doi: 10.1093/geronb/gbs069. Epub 2012 Aug 28. PMID 22929394